CLINICAL TRIAL: NCT07318025
Title: AVF-MONITOR: a New Wearable Device for Vascular Access Monitoring in Hemodialysis Patients - Proof-of-concept Study
Brief Title: AVF-MONITOR POC Proof-of-concept Study
Acronym: AVFMONITOR POC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: AVF-MONITOR POC
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Hemodyalysis
Keywords: arteriovenous fistula; hemodialysis; vascular access; monitoring; sound recording; proof-of-concept study; prototype device; vascular stenosis
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Patients undergoing HD with a functioning native AVF
  Interventions: Device: AVF MONITOR

INTERVENTIONS:
Device: AVF MONITOR — Wearable non-invasive device consisting in an electronic platform that can acquire acoustic data by means of an analog microphone.

SUMMARY:
This is a proof-of-concept single-centre prospective longitudinal interventional study performed in AVF patients under HD treatment at the Nephrology and Dialysis Department of the ASST-Papa Giovanni XXIII (Bergamo, Italy), involving the recording of AVF sounds by the AVF-MONITOR wearable prototype device.

Participants will undergo a screening and enrollment visit, then follow-up visits for AVF sounds registration will be conducted once a week for all participants, prior to dialysis session, over a period of 8 weeks.

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) is an increasingly prevalent global health issue, closely linked to the aging population. The majority of individuals with ESRD requiring renal replacement therapy undergo hemodialysis (HD) treatment . A successful HD procedure requires a well-functioning vascular access (VA) to ensure a safe and durable connection between the patient's circulation and the artificial kidney. To date, VA dysfunction remains the leading cause of morbidity and hospitalization among HD patients, representing a major limitation of this treatment modality. The current recommended VA for hemodialysis is the native arteriovenous fistula (AVF), which is surgically created in the forearm by connecting a vein and an artery through an anastomosis. Although the AVF is considered the first-choice access, it is still associated with high rates of non-maturation and early failure, with up to 40% failing within the first year post-intervention, mainly due to vascular stenosis. Identifying patients at risk of AVF failure is crucial, yet current surveillance strategies remain inadequate. In practice, AVF function is rarely monitored using the gold standard Doppler ultrasound (US) after surgical creation and initiation of HD, unless nurses report significant cannulation difficulties. By that time, however, the AVF is often already occluded, requiring the urgent placement of a central venous catheter to continue HD, followed by surgical intervention to create a new AVF. Moreover, Doppler US is time-consuming and requires a dedicated nephrologist with specific imaging expertise. Furthermore, in smaller dialysis centres, the lack of access to a Doppler US machine further restricts effective surveillance.

Continuous monitoring of AVF function could enable early identification of reduced blood flow or stenosis development, allowing timely salvage intervention by interventional radiologists before the complete closure of the AVF.

Over the years, nurses and nephrologists got used to assess AVF by palpation and auscultation, qualitatively evaluating its vibration (thrill) and the sounds it emits using a stethoscope. A non-stenotic AVF typically produces a soft, continuous murmur: a strong sound during systole and a weaker one during diastole, both associated with laminar blood flow. In contrast, a malfunctioning AVF often lacks a palpable thrill and emits a systolic-only high-pitched, hissing sound caused by turbulent and disturbed blood flow. In more severe cases of stenosis, a distinct 'whistling' sound may be heard, indicating critical dysfunction or complete failure of the AVF.

Based on these clinical evidences, recent studies have revealed significant differences in the acoustic characteristics of AVF sounds, recorded with electronic stethoscopes, between functioning and non-functioning AVFs. The frequency spectra of these sounds show that patent AVFs are characterized by low-frequency sounds, whereas stenotic AVFs exhibit higher frequencies, reaching up to 700-800 Hz. Furthermore, it has been demonstrated that AVF sounds acquired with an electronic stethoscope can be used to extract key information about hemodynamic conditions, providing indications of complex flow dynamics and adequate blood volume for effective HD. These results suggest that sound analysis has significant potential to improve clinical AVF surveillance and enhance patient outcomes.

However, the monitoring technique involving the use of an electronic stethoscope requires expert personnel, as it demands numerous precautions during both sound recording (e.g., avoiding friction and excessive pressure) and analysis, which requires technical expertise. These factors limit the use of this technological solution to only a small subset of HD patients.

To overcome these limitations, a prototype wearable device called AVF-MONITOR has been designed which allows to record AVF sound, possibly enabling simple and continuous AVF surveillance. In the future, after adequate testing, AVF-MONITOR could be potentially used in a home setting, allowing patients to independently monitor their AVF function on a daily basis.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures.
* Female and/or male aged ≥ 18.
* Patients undergoing HD with a mature and functioning native AVF.

Exclusion Criteria:

* Patients with a history of complications related to the AVF in use.
* Patients who use a graft or catheter to perform HD.
* Patients with reduced life expectancy (less than 1 year).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
High-low peak ratio | Once weekly for 8 weeks after the initial screening and enrollment visit
  Correlation between the high-low peak ratio (HLPR) calculated from acoustic recordings obtained using the AVF-MONITOR device (in Hz) and the gold standard electronic stethoscope (in Hz).

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Remuzzi, M.D., Study Director — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (1):
- ASST HPG23 - Unità di Nefrologia, Bergamo, BG, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Poloni S, Soliveri L, Caroli A, Remuzzi A, Bozzetto M. The Potential of Sound Analysis to Reveal Hemodynamic Conditions of Arteriovenous Fistulae for Hemodialysis. Ann Biomed Eng. 2025 Jan;53(1):230-240. doi: 10.1007/s10439-024-03638-2. Epub 2024 Nov 1. PMID 39485642
- [Background] Poloni S, Condemi CG, Peracchi T, Caroli A, Remuzzi A, Bozzetto M. Leveraging Acoustic Analysis to Detect Arteriovenous Fistula Complications. Kidney360. 2025 Oct 1;6(10):1771-1779. doi: 10.34067/KID.0000000840. Epub 2025 Jun 10. PMID 40493416
- [Background] Roy-Chaudhury P, Arend L, Zhang J, Krishnamoorthy M, Wang Y, Banerjee R, Samaha A, Munda R. Neointimal hyperplasia in early arteriovenous fistula failure. Am J Kidney Dis. 2007 Nov;50(5):782-90. doi: 10.1053/j.ajkd.2007.07.019. PMID 17954291
- [Background] Bozzetto M, Poloni S, Caroli A, Curto D, D'Haeninck A, Vanommeslaeghe F, Gjorgjievski N, Remuzzi A. The use of AVF.SIM system for the surgical planning of arteriovenous fistulae in routine clinical practice. J Vasc Access. 2023 Sep;24(5):1061-1068. doi: 10.1177/11297298211062695. Epub 2022 Jan 6. PMID 34986688
- [Background] Caroli A, Manini S, Antiga L, Passera K, Ene-Iordache B, Rota S, Remuzzi G, Bode A, Leermakers J, van de Vosse FN, Vanholder R, Malovrh M, Tordoir J, Remuzzi A; ARCH project Consortium. Validation of a patient-specific hemodynamic computational model for surgical planning of vascular access in hemodialysis patients. Kidney Int. 2013 Dec;84(6):1237-45. doi: 10.1038/ki.2013.188. Epub 2013 May 29. PMID 23715122
- [Background] Al-Jaishi AA, Oliver MJ, Thomas SM, Lok CE, Zhang JC, Garg AX, Kosa SD, Quinn RR, Moist LM. Patency rates of the arteriovenous fistula for hemodialysis: a systematic review and meta-analysis. Am J Kidney Dis. 2014 Mar;63(3):464-78. doi: 10.1053/j.ajkd.2013.08.023. Epub 2013 Oct 30. PMID 24183112